CLINICAL TRIAL: NCT06986382
Title: Phase 1b/2a Trial of Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) From an HLA-partially Matched Related or Unrelated Donor After TCRab+ T-cell/CD19+ B-cell Depletion for Patients With Monogenic and/or Early-onset (EO), Medically Refractory (MR) Crohn Disease (CD)
Brief Title: Phase 1b/2a Trial of Allogeneic HSCT From an HLA-partially Matched Related or Unrelated Donor After TCRab+ T-cell/CD19+ B-cell Depletion for Patients With Monogenic and/or Early-onset Medically Refractory Crohn Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jessie L. Alexander, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78920
Record Dates: First submitted 2025-05-20; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Prednisone; Fibroblast Growth Factor 7; Clofarabine; Melphalan; Whole-Body Irradiation; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cohort 1b: Safety Lead-In (Experimental): An initial cohort of 4 patients will be enrolled as part of the initial Phase 1b safety run-in evaluation. Patients will undergo an αβdepleted hematopoietic stem cell transplant (HSCT) after receiving a conditioning regimen.
  Interventions: Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System; Drug: Prednisone/Methylprenisolone; Drug: Palifermin; Drug: ATG; Drug: Clofarabine; Drug: Melphalan; Radiation: Total Body Irradiation; Drug: Rituximab
- Cohort 2a (Experimental): If the intervention is determined to be safe and non-futile, the study will continue to enroll 10 more patients under Phase 2a following the same treatment as Phase 1b.
  Interventions: Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System; Drug: Prednisone/Methylprenisolone; Drug: Palifermin; Drug: ATG; Drug: Clofarabine; Drug: Melphalan; Radiation: Total Body Irradiation; Drug: Rituximab

INTERVENTIONS:
Device: CliniMACS® TCR α/β Reagent Kit and CliniMACS® CD19 System — CliniMACS® TCRαβ-Biotin and CD19 Systems will be used to create the mobilized peripheral blood stem cells (PBSC) from allogeneic donors depleted of TCRαβ+ T cells and CD19+ B cells to be infused into the patient for the HSCT. The target dose for the number of CD34+ HSC infused is > 10 x 10^6 cells/Kg recipient weight. The minimum dose is 2 x 10^6 cells/Kg. There is no upper limit to the dose of CD34+ HSC infused as long as no more than 1 x 10^5 TCRαβ+ T-cells/Kg are infused. The target dose of TCRαβ+ T cells/Kg is < 0.50 x 10^5.
  Other Names: TCRαβ+ T-cells
Drug: Prednisone/Methylprenisolone — Administered as part of the HSCT conditioning regimen
Drug: Palifermin — Administered as part of the HSCT conditioning regimen
Drug: ATG — Administered as part of the HSCT conditioning regimen
Drug: Clofarabine — Administered as part of the HSCT conditioning regimen
Drug: Melphalan — Administered as part of the HSCT conditioning regimen
Radiation: Total Body Irradiation — 200 cGy, administered as part of the HSCT conditioning regimen
Drug: Rituximab — Administered as part of the HSCT conditioning regimen

SUMMARY:
This research study is investigating whether alpha beta T-cell depleted hematopoietic stem cell transplant (HSCT) can be an immune system replacement for Crohn disease patients and whether this is safe and effective for patients with early onset, medically refractory Crohn disease.

DETAILED DESCRIPTION:
This is a single center, non-randomized, non-controlled open-label Phase 1b/2a trial to study the safety and efficacy of performing TCRαβ+ T-cell/CD19+ B-cell depleted (TCRαβ-depleted) HSCT to induce immune tolerance in patients with monogenic or early onset, medically refractory Crohn disease to re-establish normal immune-intestinal homeostasis.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Meets at least one of the following criteria:

a. Known monogenic ("Mendelian") cause of IBD for which HSCT has been successfully performed i. Causative gene mutation known for which HSCT is demonstrated to be curative (e.g., IL10, IL10RA, IL10RB, XIAP, IPEX, WAS, CD40L, CGD, LRBA, CTLA4, DOCK8 and SCID syndromes).

b. Known monogenic cause of CD for which HSCT has not been previously performed i. Causative gene mutation expressed in lymphohematopoietic cells, for which HSCT has not been previously performed; AND ii. Moderate disease activity (shown through endoscopic, MRI, or PCDAI score); AND iii. Has been treated with at least two available treatment pathways (e.g., TNF inhibitors, anti-IL12 and /or IL-23 antibodies, JAK inhibitors, anti-integrin), but did not have adequate response, experienced significant toxicity, or had adverse effect(s) c. Suspected monogenic cause of CD i. Rare variant in a gene predicted to be functionally deleterious, suspected to drive IBD, and expressed in lymphohematopoietic cells; AND ii. Moderate disease activity or corticosteroid-dependence despite trials of at least two biologic or small molecule therapies of different mechanisms or significant toxicity or adverse effect related to such medical therapy.

d. Medically refractory CD with suspected strong genetic component, but no clearly identified deleterious single gene mutation.

i. Moderate or severe disease activity with either:

1. history of corticosteroid-dependence despite trials of at least two biologic or small molecule therapies of different mechanisms,
2. significant toxicity, or adverse effects related to such medical therapy;

AND at least one of the following criteria from ii or iii below:

ii. Severity unlikely to be tolerable long-term due to the presence of either:

1. Disease not amenable to surgical therapy without risk of short bowel syndrome or permanent ileostomy;
2. Requirement for long-term parenteral nutrition;
3. Intolerable extraintestinal symptoms (e.g., arthritis, dermatitis); iii. Presence of any of the following features associated with high genetic contribution to disease:

1. Parental consanguinity 2. Strong family history of IBD (present in first degree relatives) 3. Diagnosis earlier than 6 years of age 4. Extraintestinal manifestations 5. Family history of CD, IBD or autoimmune disease 2. Age >2 year and < 30 years. 3. The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DQB1 and HLA-DRB1.

4. Lansky/Karnofsky score ≥50; the Karnofsky Scale will be used in subjects ≥ 16 years of age, and the Lansky Scale will be used for those < 16 years of age.

5. All subjects ≥ 18 years of age must be able to give informed consent, or adults lacking capacity to consent must have a legally authorized representative (LAR) available to provide consent. For subjects <18 years old their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric subjects will be included in age-appropriate discussion and written assent will be obtained for those > 7 years of age, when appropriate.

6. Female subjects of childbearing potential must agree to use an effective means of birth control to avoid pregnancy throughout the transplant procedure, while on immunosuppression.

Recipient Exclusion Criteria:

1. Ulcerative colitis
2. CD and associated extraintestinal manifestations responsive to medical therapy without corticosteroid-dependence or significant toxicity or adverse effects
3. Known or suspected functionally deleterious mutation in a gene that meets either of the following expression criteria:

   1. Specifically expressed in epithelial or stromal cells, but not expressed in lymphohematopoietic cells (e.g., TTC7A)
   2. Expected to be more functionally deleterious in cell types other than lymphohematopoietic cells than in lymphohematopoietic cell types
4. Active hemophagocytic lymphohistiocytosis (HLH). Patients with a history of hemophagocytic lymphohistiocytosis (HLH) are eligible, if there is no current clinical, histological, or biochemical evidence of HLH activity.
5. Dysfunction of liver, defined as:

   1. ALT/AST > 5 times upper normal value, or direct bilirubin > 3 times upper normal value; or
   2. Cirrhosis with bridging fibrosis (grade F3 or greater) or sclerosing cholangitis
6. Severe cardiovascular disease (e.g. left ventricular ejection fraction < 40%), or clinical or echocardiographic evidence of severe diastolic dysfunction.
7. Severe renal dysfunction defined as serum creatinine >1.5 X upper limit of normal (ULN) or 24-hour creatinine clearance <50 ml/min/m2
8. Human immunodeficiency virus (HIV)-infected patients or patients with evidence of chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
9. Past exposure to therapeutic radiation.
10. Previous allogeneic HSCT. Patients who have received previous autologous HSCT are eligible.
11. Active malignancy and patients who have history of malignancies, unless disease free for at least 2 years, with the exception of nonmelanoma skin cancer or carcinoma in situ (e.g., bladder, breast).
12. Pregnant or lactating females.
13. Lack of patient/parent/guardian informed consent.
14. Any severe concurrent uncontrolled disease which, in the judgement of the investigator, would place the patient at increased risk during participation in the study, other than primary disease.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2037-07 (Estimated); Study Completion 2040-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with myeloid engraftment | Day 42 post-HSCT
  Cumulative incidence of donor myeloid engraftment by Day +42 post-HSCT. Myeloid engraftment is defined as ANC of > 0.5 x 109/L for three consecutive laboratory values obtained on different days. Date of myeloid engraftment is the first date of the three lab values taken.
Number of patients with Grade III-IV acute graft vs host disease (GVHD) | Day 90 and 180 post-HSCT
  Cumulative incidence of acute GvHD (graded as II-IV and III-IV using the Magic criteria)
  Cumulative incidence of acute GvHD (graded as II-IV and III-IV using the Magic criteria)
  Cumulative incidence of acute GvHD (graded as II-IV and III-IV using the Magic criteria)
  Cumulative incidence of acute GvHD (graded using the Magic criteria)
Number of patients in remission of Crohn disease (Calprotectin) | 2 years post-HSCT
  Cumulative incidence of patient who achieve remission defined by fecal calprotectin values less than 250 mg/g
Number of patients in remission of Crohn disease (wPCDAI or CDAI) | 2 years post-HSCT
  Cumulative incidence of remission demonstrated by weighted Pediatric Crohn's Disease Activity Index (wPCDAI) <12.5 or Crohn's Disease Activity Index (CDAI) of <150 if adult

SECONDARY OUTCOMES:
Number of patients who achieve normal immune function derived from donor cells | 1 year post-HSCT
  Cumulative incidence of patients with age-appropriate normalization of peripheral blood lymphocyte numbers including T, NK and B cells
Number of patients who achieve full donor chimerism | 1 year post-HSCT
  Cumulative incidence of patient chimerism defined as >95% of donor cells as assessed by peripheral blood (total, CD15+, CD3+, CD56+, CD19+, and CD34+) chimerism by short tandem repeat (STR) or next generation sequencing (NGS) analysis
Number of patients with healthy immune cell function | 1 year post-HSCT
  Cumulative incidence of patients who have mitogen and antigen specific T-cell proliferation or cytokine release in response to in vitro stimulation
Number of patients who regain CD3 cells | Day 90 and 180 post-HSCT
  CD3 cell count of >200/ uL
Number of patients who experience moderate and severe chronic GvHD | 1 year post-HSCT
  Cumulative incidence of patients experiencing moderate or severe chronic GvHD by NIH Consensus Criteria for Organ scoring of cGVHD
Number of patients who experience severe infections | 1 year post-HSCT
  Cumulative incidence of patients experiencing Grade 3 or higher CTCAE infections after HSCT
Patient survival | 2 and 5 years post-HSCT
Number of patients with response in Crohn disease activity - 50% CRP or higher | 1 and 2 years post-HSCT
  Cumulative incidence of patients who have a <0.5 mg/dL reduction in C-reactive protein (CRP)
Number of patients with response in Crohn disease activity - wPCDAI/CDAI | 1 year post-HSCT
  Cumulative incidence of patients who achieve wPCDAI score reduced by 17.5 points from baseline if pediatric, CDAI reduced by at least 100 points from baseline if adult
Number of patients with endoscopic healing | 2 years post-HSCT
  Endoscopic healing defined as ≤1 SEMA score
Number of patients with sustained steroid-free remission | 2 years post-HSCT
  Cumulative incidence of patients who are able to discontinue steroids for 3 or more months

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Alexander, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kammermeier J, Dziubak R, Pescarin M, Drury S, Godwin H, Reeve K, Chadokufa S, Huggett B, Sider S, James C, Acton N, Cernat E, Gasparetto M, Noble-Jamieson G, Kiparissi F, Elawad M, Beales PL, Sebire NJ, Gilmour K, Uhlig HH, Bacchelli C, Shah N. Phenotypic and Genotypic Characterisation of Inflammatory Bowel Disease Presenting Before the Age of 2 years. J Crohns Colitis. 2017 Jan;11(1):60-69. doi: 10.1093/ecco-jcc/jjw118. Epub 2016 Jun 14. PMID 27302973
- [Background] de Lange KM, Moutsianas L, Lee JC, Lamb CA, Luo Y, Kennedy NA, Jostins L, Rice DL, Gutierrez-Achury J, Ji SG, Heap G, Nimmo ER, Edwards C, Henderson P, Mowat C, Sanderson J, Satsangi J, Simmons A, Wilson DC, Tremelling M, Hart A, Mathew CG, Newman WG, Parkes M, Lees CW, Uhlig H, Hawkey C, Prescott NJ, Ahmad T, Mansfield JC, Anderson CA, Barrett JC. Genome-wide association study implicates immune activation of multiple integrin genes in inflammatory bowel disease. Nat Genet. 2017 Feb;49(2):256-261. doi: 10.1038/ng.3760. Epub 2017 Jan 9. PMID 28067908
- [Background] Graham DB, Xavier RJ. Pathway paradigms revealed from the genetics of inflammatory bowel disease. Nature. 2020 Feb;578(7796):527-539. doi: 10.1038/s41586-020-2025-2. Epub 2020 Feb 26. PMID 32103191
- [Background] Crowley E, Warner N, Pan J, Khalouei S, Elkadri A, Fiedler K, Foong J, Turinsky AL, Bronte-Tinkew D, Zhang S, Hu J, Tian D, Li D, Horowitz J, Siddiqui I, Upton J, Roifman CM, Church PC, Wall DA, Ramani AK, Kotlarz D, Klein C, Uhlig H, Snapper SB, Gonzaga-Jauregui C, Paterson AD, McGovern DPB, Brudno M, Walters TD, Griffiths AM, Muise AM. Prevalence and Clinical Features of Inflammatory Bowel Diseases Associated With Monogenic Variants, Identified by Whole-Exome Sequencing in 1000 Children at a Single Center. Gastroenterology. 2020 Jun;158(8):2208-2220. doi: 10.1053/j.gastro.2020.02.023. Epub 2020 Feb 19. PMID 32084423
- [Background] Cifaldi C, Chiriaco M, Di Matteo G, Di Cesare S, Alessia S, De Angelis P, Rea F, Angelino G, Pastore M, Ferradini V, Pagliara D, Cancrini C, Rossi P, Bertaina A, Finocchi A. Novel X-Linked Inhibitor of Apoptosis Mutation in Very Early-Onset Inflammatory Bowel Disease Child Successfully Treated with HLA-Haploidentical Hemapoietic Stem Cells Transplant after Removal of alphabeta+ T and B Cells. Front Immunol. 2017 Dec 22;8:1893. doi: 10.3389/fimmu.2017.01893. eCollection 2017. PMID 29312354
- [Background] Stiff PJ, Leinonen M, Kullenberg T, Rudebeck M, de Chateau M, Spielberger R. Long-Term Safety Outcomes in Patients with Hematological Malignancies Undergoing Autologous Hematopoietic Stem Cell Transplantation Treated with Palifermin to Prevent Oral Mucositis. Biol Blood Marrow Transplant. 2016 Jan;22(1):164-9. doi: 10.1016/j.bbmt.2015.08.018. Epub 2015 Aug 22. PMID 26303102
- [Background] Alatrash G, Thall PF, Valdez BC, Fox PS, Ning J, Garber HR, Janbey S, Worth LL, Popat U, Hosing C, Alousi AM, Kebriaei P, Shpall EJ, Jones RB, de Lima M, Rondon G, Chen J, Champlin RE, Andersson BS. Long-Term Outcomes after Treatment with Clofarabine +/- Fludarabine with Once-Daily Intravenous Busulfan as Pretransplant Conditioning Therapy for Advanced Myeloid Leukemia and Myelodysplastic Syndrome. Biol Blood Marrow Transplant. 2016 Oct;22(10):1792-1800. doi: 10.1016/j.bbmt.2016.06.023. Epub 2016 Jul 1. PMID 27377901
- [Background] Bertaina A, Grimm PC, Weinberg K, Parkman R, Kristovich KM, Barbarito G, Lippner E, Dhamdhere G, Ramachandran V, Spatz JM, Fathallah-Shaykh S, Atkinson TP, Al-Uzri A, Aubert G, van der Elst K, Green SG, Agarwal R, Slepicka PF, Shah AJ, Roncarolo MG, Gallo A, Concepcion W, Lewis DB. Sequential Stem Cell-Kidney Transplantation in Schimke Immuno-osseous Dysplasia. N Engl J Med. 2022 Jun 16;386(24):2295-2302. doi: 10.1056/NEJMoa2117028. PMID 35704481
- [Background] Greco R, Labopin M, Badoglio M, Veys P, Furtado Silva JM, Abinun M, Gualandi F, Bornhauser M, Ciceri F, Saccardi R, Lankester A, Alexander T, Gennery AR, Bader P, Farge D, Snowden JA. Allogeneic HSCT for Autoimmune Diseases: A Retrospective Study From the EBMT ADWP, IEWP, and PDWP Working Parties. Front Immunol. 2019 Jul 4;10:1570. doi: 10.3389/fimmu.2019.01570. eCollection 2019. PMID 31333680
- [Background] McLaughlin L, DeZoeten E, Verneris MR. Can allogeneic haematopoietic cell transplantation be curative in classical Crohn's disease? Br J Haematol. 2023 Mar;200(5):541-542. doi: 10.1111/bjh.18551. Epub 2022 Nov 9. PMID 36352551
- [Background] Moser LM, Fekadu J, Willasch A, Rettinger E, Sorensen J, Jarisch A, Kirwil M, Lieb A, Holzinger D, Calaminus G, Bader P, Bakhtiar S. Treatment of inborn errors of immunity patients with inflammatory bowel disease phenotype by allogeneic stem cell transplantation. Br J Haematol. 2023 Mar;200(5):595-607. doi: 10.1111/bjh.18497. Epub 2022 Oct 10. PMID 36214981
- [Background] Engelhardt KR, Shah N, Faizura-Yeop I, Kocacik Uygun DF, Frede N, Muise AM, Shteyer E, Filiz S, Chee R, Elawad M, Hartmann B, Arkwright PD, Dvorak C, Klein C, Puck JM, Grimbacher B, Glocker EO. Clinical outcome in IL-10- and IL-10 receptor-deficient patients with or without hematopoietic stem cell transplantation. J Allergy Clin Immunol. 2013 Mar;131(3):825-30. doi: 10.1016/j.jaci.2012.09.025. Epub 2012 Nov 14. PMID 23158016
- [Background] Lopez-Cubero SO, Sullivan KM, McDonald GB. Course of Crohn's disease after allogeneic marrow transplantation. Gastroenterology. 1998 Mar;114(3):433-40. doi: 10.1016/s0016-5085(98)70525-6. PMID 9496932